CLINICAL TRIAL: NCT04024813
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled, Multiple Center Study to Evaluate the Safety, Tolerability, and Efficacy of Seladelpar Administered for 24 Weeks in Adult Patients With Primary Sclerosing Cholangitis (PSC)
Brief Title: A Study to Evaluate the Safety, and Tolerability, and Efficacy of Seladelpar in Patients With PSC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated as a precautionary measure due to histological findings in a nonalcoholic steatohepatitis (NASH) study (CB8025-21730, NCT03551522).
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB8025-21845; 2019-001760-30 (EudraCT Number)
Record Dates: First submitted 2019-06-20; First posted 2019-07-18 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC; Cholangitis, Sclerosing; Cholangitis; Bile Duct Diseases; Biliary Tract Diseases; Digestive System Diseases
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangitis; Bile Duct Diseases; Biliary Tract Diseases; Digestive System Diseases | interventions — seladelpar; (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Dose masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (N=25) (Placebo Comparator): Placebo for the remainder of the study
  Interventions: Drug: Placebo to match Seladelpar
- Seladelpar 5 mg (N=25) (Experimental): 5 mg seladelpar daily for the remainder of the study
  Interventions: Drug: Seladelpar
- Seladelpar 10 mg (N=25) (Experimental): 10 mg seladelpar for the remainder of the study
  Interventions: Drug: Seladelpar
- Seladepar 25 mg (N=25) (Experimental): 25 mg seladelpar for the remainder of the study
  Interventions: Drug: Seladelpar

INTERVENTIONS:
Drug: Seladelpar — Capsule(s) administered orally once daily
  Other Names: MBX-8025; Livdelzi®
  Arms: Seladelpar 10 mg (N=25); Seladelpar 5 mg (N=25); Seladepar 25 mg (N=25)
Drug: Placebo to match Seladelpar — Capsule(s) administered orally once daily
  Arms: Placebo (N=25)

SUMMARY:
The objectives of this study are to evaluate the effect of seladelpar treatment compared to placebo on efficacy, safety, and tolerability in patients with primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of primary sclerosing cholangitis (PSC) based on any two of the following three criteria:

   * Historical evidence of an elevated alkaline phosphatase (AP) > upper limit of normal (ULN) from any prior laboratory result
   * Liver biopsy consistent with PSC
   * Abnormal cholangiography consistent with PSC as measured by magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography (ERCP), or percutaneous transhepatic cholangiography (PTC)
2. Individuals must have the following specific additional laboratory parameters measured by the Central Laboratory at Screening:

   * AP ≥ 1.5 × ULN and < 8 × ULN
   * Total bilirubin ≤ 2 × ULN
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN
   * Estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73 m^2
   * Platelets ≥ 140 × 10^3/µL
   * International Normalized Ratio (INR) ≤ 1.3 (in the absence of warfarin or other anticoagulant therapy)
   * Albumin ≥ 3.5 g/dL
3. Patients taking ursodeoxycholic acid (UDCA) will be allowed to enroll if meeting the following criteria:

   * Total daily dose of ≤ 20 mg/kg/day
   * A minimum of 6 months of stable treatment
   * Minimum of 12 weeks off treatment prior to Screening if UDCA is recently discontinued

Key Exclusion Criteria:

1. Clinically significant acute or chronic liver disease of an etiology other than PSC
2. Patients with a diagnosis of overlapping autoimmune hepatitis (AIH) and PSC
3. Secondary or immunoglobulin G4 (IgG4) related sclerosing cholangitis
4. Small duct PSC
5. Presence of a cholangiocarcinoma on cholangiography or MRI at Screening as determined by the central radiologist and the principal investigator (PI) or medical monitor
6. Bile duct stent or percutaneous bile duct drain placement, or balloon dilatation procedure of a stricture within 12 weeks of Screening
7. History, evidence, or high suspicion of cholangiocarcinoma or other hepatobiliary malignancy based on imaging, screening laboratory values, and/or clinical symptoms
8. Presumptive or diagnosed acute cholangitis within 12 weeks of Screening and through Day 1
9. Evidence of compensated or decompensated cirrhosis based on histology, relevant medical complications, or laboratory parameters:

   * Historical liver biopsy demonstrating cirrhosis (eg, Ludwig Stage 4 or Ishak Stage 5)
   * Current or prior history of decompensated liver disease, including ascites, hepatic encephalopathy, variceal bleeding or other clinical conditions consistent with cirrhosis and/or portal hypertension,
   * Liver stiffness > 14.4 kPa by FibroScan, or
   * Combined low platelet count (< 140 × 10^3/µL ) with one of the following:

     * Serum albumin < 3.5 g/dL,
     * INR > 1.3 (not due to antithrombotic agent use), or
     * Total bilirubin > ULN
10. Prior or actively listed for liver transplantation
11. Prior exposure to seladelpar

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (10):
- United States (8):
  - Sutter Pacific Medical Foundation - California Pacific Medical Center, San Francisco, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Henry Ford Health System, Novi, Michigan
  - New York University, New York, New York
  - Liver Institute of Virginia, Newport News, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
- Toronto Centre for Liver Disease-Toronto General Hospital, Toronto, Ontario, Canada
- ID Clinic, Mysłowice, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was to be conducted in 60 sites in Australia, Europe, Israel, and North America. Only 1 site in the United States enrolled. The study was terminated early and only 1 participant was enrolled in the placebo arm.
Groups:
- Placebo: Participant received placebo once daily until Day 14.
Period: Overall Study
Arm/Group | Placebo
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Placebo
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  65 to 84 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Baseline Serum Alkaline Phosphatase (AP) at Week 24
Time Frame: Baseline, Week 24
Population: The study was terminated before the outcome measure data were collected.
Arm/Group | Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were planned to be collected up to 24 weeks. Due to the early study termination, data is reported up to Day 59.
Time Frame: Up to Day 59
Population: The data for the participant that enrolled and received placebo was included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Incidence of Primary Sclerosing Cholangitis (PSC)-Related Symptoms or Procedures
Time Frame: Up to 24 weeks
Population: The study was terminated before the outcome measure data were collected.
Arm/Group | Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Hepatic Disease Progression Events
Description: Hepatic disease progression events is defined by the first occurrence of the following events: liver transplantation, Model for End-Stage Liver Disease (MELD) score ≥ 15, hepatic decompensation events, and hepatocellular carcinoma.
Time Frame: Up to 24 weeks
Population: The study was terminated before the outcome measure data were collected.
Arm/Group | Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Day 59
Description: The data for the participant that enrolled and received placebo was included.
Arm/Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated early and only 1 participant enrolled in the placebo arm and received placebo up to Day 14. The pre-specified analyses were not conducted due to study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT04024813/Prot_SAP_001.pdf